CLINICAL TRIAL: NCT06605768
Title: A 3-Month, Randomized, Single-Blind, Placebo-Controlled Study Evaluating the Ability of Nutra Harmony "Biotin, Collagen &Amp;Amp; Keratin Beauty Complex" Dietary Supplement Promotion in Hair Thickness and Hair Strength in Individuals With Self-Perceived Thinning Hair
Brief Title: Study Evaluating the Effects of Dietary Supplement on Hair Thickness and Hair Strength in Individuals With Self-Perceived Thinning Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutra Harmony LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nutra 1-0602
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Hair Thinning
Keywords: Hair thinning; hair thickness; hair strength; hair falling; women; oral supplement
MeSH Terms: conditions — Alopecia | interventions — Biotin; Collagen; Keratins; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo product
- Group Treatment (Active Comparator)
  Interventions: Dietary Supplement: Complex with Biotin, Collagen, Keratin, Hyaluronic Acid.

INTERVENTIONS:
Dietary Supplement: Complex with Biotin, Collagen, Keratin, Hyaluronic Acid. — Biotin, Collagen & Keratin Beauty Complex" 30,000 mcg, 60 capsules, oral route of administration.
  Arms: Group Treatment
Dietary Supplement: Placebo product — Placebo, 60 capsules, oral route of administration
  Arms: Group Placebo

SUMMARY:
The Nutra Harmony "Biotin, Collagen & Keratin Beauty Complex" is an oral food/dietary supplement specifically designed to promote hair growth for people suffering from temporary thinning hair. The hypothesis of this clinical research study is that the ingestion of "Biotin, Collagen & Keratin Beauty Complex" for over a three (3) month period will strengthen the hair and increase hair thickness by promoting the growth of terminal hairs in subjects, ages 21-50 years of age with self-perceived thinning hair associated with poor diet, stress, hormonal influences when compared to using the placebo tablet.

DETAILED DESCRIPTION:
This study was a two-arm, parallel group, double-blind, placebo-controlled trial powered to detect meaningful differences in the hair growth for people suffering from temporary thinning hair between the treatment(main) and control groups at 3 months. Participants of the main group were prescribed the "Biotin, Collagen & Keratin Beauty Complex" 30,000 mcg, 60 capsules produced by NUTRA HARMONY LLC, participants of the control group were prescribed placebo (microcrystalline cellulose (MCC)), 60 capsules manufactured by NUTRA HARMONY LLC. The duration of study in both groups of subjects was 3 months and the treatment period continued for 90 days following randomization. A total of 80 males and females aged 21 to 50 with temporary thinning hair who meet all eligibility criteria were randomized in this study. Within the study, there were a total of 6 site visits for each participant, during which the following procedures were performed:

Visit 1 (Screening visit):

Signing the informed consent document Demography recording Height, weight assessment Vital signs: pulse, systolic [SBP] and diastolic [DBP] blood pressure, after 10 minutes of resting position Medical history & Current medications Hematology A urine pregnancy test (for women of childbearing potential Physical examination: general/appearance; head, eyes, ears, nose, throat, and oropharynx; skin evaluations; respiratory; cardiovascular; abdomen/gastrointestinal; urological system, musculoskeletal system and neurological system High-quality clinical and dermoscopic photographs of hair in the target area of the scalp made by dermatoscope High-quality photographs of hair in the target area of the scalp made by digital camera Quality of Life Questionnaire

Visit 2 (Randomization):

Vital signs: pulse, systolic [SBP] and diastolic [DBP] blood pressure, after 10 minutes of resting position Study Intervention randomization: participants will be assigned randomly in a 1:1 ratio to study product or placebo.

Visit 3 (Day 21), Visit 4 (Day 40), Visit 5 (Day 60):

Vital signs: pulse, systolic [SBP] and diastolic [DBP] blood pressure, after 10 minutes of resting position Counting the amount of hair that fell out with each wash Determining the change in hair area compared to the baseline Counting the amount of hair in several control points compared to the baseline

Visit 6 (Day 90, End of Study):

Vital signs: pulse, systolic [SBP] and diastolic [DBP] blood pressure, after 10 minutes of resting position Hematology Counting the amount of hair that fell out with each wash Determining the change in hair area compared to the baseline Counting the amount of hair in several control points compared to the baseline High-quality clinical and dermoscopic photographs of hair in the target area of the scalp made by dermatoscope High-quality photographs of hair in the target area of the scalp made by digital camera Quality of Life Questionnaire Self-assessment Questionnaire

The effectiveness of the treatment was evaluated by considering the increase in hair growth in study supplement-treated subjects, which was defined by determining the change in hair area from the baseline and counting the amount of hair in several control points from the baseline comparing to placebo-treated subjects, as well as hair washing (shampooing) for hair shedding counts in study supplement-treated subjects comparing to placebo-treated subjects and the change in patient quality of life questionnaires and self-assessment questionnaires during and following the study.

The tolerability of the studied supplement was assessed on the basis of the patient's subjective complaints, the presence and severity of adverse reactions/side effects, the data of the patient's examination and laboratory examination.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals, ages 21-50 years of age.
2. Clinically-determined general good health as determined by responses to the initial study assessment.
3. Individuals with self-perceived thinning hair associated with poor diet, stress, hormone influences.
4. Individuals willing to maintain their normal hair shampooing frequency.
5. Individuals willing to add the provided oral supplement to their current daily routine.
6. Individuals willing to not substantially change their current diet, medications, or exercise routines for the duration of the study. If a subject receives physician guidance during the study to change diet, medications, or exercise routine, the subject will need to notify the clinic as soon as possible.
7. Individuals willing to undergo a physical exam to include height, weight, blood pressure, pulse, general physical findings, scalp exam and blood sample collection.
8. Individuals with Fitzpatrick I-IV photo skin types.
9. Willingness to have digital photography of the target area and scalp for hair counts at Visits 1, 2, 3, 4, 5, 6.
10. Willingness to have their hair washed (shampooed) over a sink containing cheesecloth for hair shedding counts at Visit 1, 2, 3, 4, 5, 6.
11. Willingness to maintain a consistent haircut and hair color throughout the 3-months study period and to come to visits with clean (shampoo must be done 24 hours or more prior to the visit) and dry hair.
12. Willingness of subjects who have color treated hair to have the color treatment performed at the same time interval prior to each visit (i.e. If on Visit 1 the color treatment was done one week prior then the color treatment is expected to occur at a similar interval of one week prior to Visit 2, 3 ,4 ,5, 6).
13. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Individuals with a known history of intolerance or allergy to fish, seafood/shellfish or acerola.
2. Individuals with any known allergy or sensitivity to any shampoo/conditioner.
3. Females who are nursing, pregnant, planning to become pregnant during the study.
4. Individuals with known stressful incident within the last six months (i.e. death in family, miscarriage).
5. Individuals who are participating on any clinical research study at another research center or doctor's office.
6. Females who have recently (within the last 6 months) started the use of hormones for birth control or hormone replacement therapy (HRT). Women currently using hormones for birth control or HRT must have been on a stable dose (6 months or longer) in order to be eligible for the study.
7. Individuals currently using light therapy to treat thinning hair.
8. Individuals who have regularly used Rogaine (Minoxidil) within the last 3 months.
9. Individuals currently using any other biotin/keratin/collagen supplements.
10. Individuals who have used prescription drugs known to affect the hair growth cycle within the last 6 months (e.g., hormone-based birth control for less than 6 months, cyproterone acetate, Aldactone/spironolactone, Finasteride or any 5-alpha-reductase inhibitor).
11. Individuals suffering from other hair loss disorders, such as alopecia areata, scarring alopecia, androgenetic alopecia and telogen effluvium as determined on initial study assessment by the Investigator.
12. Individuals with self-reported uncontrolled diseases (i.e. diabetes, hypertension, hyperthyroidism, hypothyroidism, etc.). Medical conditions that are under control with or without treatment will be considered on an individual basis by the Investigators.
13. Individuals with self-reported active hepatitis, immune deficiency, HIV or autoimmune disease.
14. Individuals having a known active dermatologic condition which, in the opinion of the examining Investigators, might place the subject at a greater risk or interfere with clinical evaluations (e.g., seborrheic dermatitis, psoriasis, atopic dermatitis, advanced skin cancer, etc.).

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Limited Liability Company Treatment and Diagnostic Center ADONIS Plus, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No
IPD (Individual Participant Data) will not be shared, as information about each participant is strictly confidential. Only aggregated information regarding the effectiveness and safety of the investigated supplement among all study participants will be shared within the framework of statistical data.

REFERENCES:
- [Background] Thom E. Efficacy and tolerability of Hairgain in individuals with hair loss: a placebo-controlled, double-blind study. J Int Med Res. 2001 Jan-Feb;29(1):2-6. doi: 10.1177/147323000102900101. PMID 11277343
- [Background] Williamson D, Gonzalez M, Finlay AY. The effect of hair loss on quality of life. J Eur Acad Dermatol Venereol. 2001 Mar;15(2):137-9. doi: 10.1046/j.1468-3083.2001.00229.x. PMID 11495520

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single outpatient research center (ADONIS Plus, Kyiv, Ukraine). Enrollment began on 19 Feb 2024 (first informed consent). Participants attended a site screening visit and, if eligible, were randomized and assigned to supplement or placebo. Study procedures continued through 12 Jul 2024 (last study procedure).
Pre-assignment Details: None. After completion of screening assessments, eligible participants were randomized and assigned to supplement or placebo on the same day (no washout or run-in period).
Groups:
- Group Placebo: Participants received matching placebo capsules containing microcrystalline cellulose (MCC). Dosing: 1 capsule orally twice daily for 90 days (from Visit 2/Day 1 through Visit 6/Day 90).
- Group Treatment: Participants received the investigational product "Biotin, Collagen & Keratin Beauty Complex" oral capsules. Dosing: 1 capsule orally twice daily for 90 days (from Visit 2/Day 1 through Visit 6/Day 90).
Period: Overall Study
Arm/Group | Group Placebo | Group Treatment
Started | 40 | 40
Completed | 39 | 38
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for participants included in the baseline summary table (Treatment n=40; Placebo n=37).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group Placebo | Group Treatment | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Customized [Count of Participants; unit: Participants] — Age categories at baseline (years).
  Participants
    21-30 | 13 | 9 | 22
    31-40 | 10 | 16 | 26
    41-50 | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants] — Sex at baseline.
  Participants
    Female | 30 | 37 | 67
    Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hair Shedding (1-2 hair per unit) [Count of Participants; unit: Participants] — Hair shedding at baseline was assessed by trichoscopic examination as the presence of 1-2 shed hairs per follicular unit (hair unit) in the examined scalp area. Results are reported as the number of participants meeting this criterion at baseline in each study group.
  Participants | 27 | 24 | 51
Hair thinning [Count of Participants; unit: Participants] — Hair thinning at baseline was evaluated clinically and/or by trichoscopy as visible reduction in hair shaft caliber and/or overall decreased hair density in the examined scalp area. Results are reported as the number of participants with hair thinning present at baseline in each study group.
  Participants | 18 | 20 | 38
Increase in the amount of vellus hair compared to mature hairs [Count of Participants; unit: Participants] — At baseline, the proportion of vellus hairs relative to mature (terminal) hairs was assessed by trichoscopy in the examined scalp area. An increased amount of vellus hair compared with mature hairs was recorded when vellus hairs predominated relative to mature hairs. Results are reported as the number of participants meeting this criterion at baseline in each study group.
  Participants | 10 | 10 | 20
Increased distance between units [Count of Participants; unit: Participants] — Increased distance between follicular units at baseline was assessed by trichoscopy as widened spacing between hair units in the examined scalp area, consistent with reduced hair density. Results are reported as the number of participants with increased inter-unit distance present at baseline in each study group.
  Participants | 14 | 13 | 27
Inflammatory processes in the scalp and blood vessels [Count of Participants; unit: Participants] — Signs of inflammatory processes in the scalp and scalp blood vessels at baseline were assessed by clinical examination and/or trichoscopy (e.g., erythema, perifollicular inflammation, and/or vascular/inflammatory changes). Results are reported as the number of participants with inflammatory findings present at baseline in each study group.
  Participants | 15 | 23 | 38

OUTCOME MEASURES:

1. Primary Outcome: Hair Shedding (1-2 Hairs Per Unit)
Description: Hair shedding was assessed by trichoscopic evaluation of the target scalp area. The endpoint reflects the proportion of participants meeting the criterion of 1-2 shed hairs per follicular unit at the specified time point.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Group Placebo | Group Treatment
Number analyzed (Participants) | 39 | 38
Participants
  Shedding not present | 21 | 10

2. Secondary Outcome: Hair Thinning
Description: Hair thinning was evaluated in the target scalp area using standardized trichoscopic assessment. The endpoint reflects the proportion of participants with visible hair shaft thinning/decreased hair caliber at the specified time point.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Group Placebo | Group Treatment
Number analyzed (Participants) | 39 | 38
Participants | 17 | 7

3. Secondary Outcome: Increase in the Amount of Vellus Hair Compared to Mature Hairs
Description: The vellus-to-terminal hair pattern was assessed by trichoscopy in the target scalp area. The endpoint reflects the proportion of participants with an increased proportion of vellus hairs compared with mature (terminal) hairs at the specified time point.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Group Placebo | Group Treatment
Number analyzed (Participants) | 39 | 38
Participants | 14 | 22

4. Secondary Outcome: Increased Distance Between Units
Description: Inter-unit spacing was assessed by trichoscopy in the target scalp area. The endpoint reflects the proportion of participants with an increased distance between follicular units, indicating reduced follicular density, at the specified time point.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Group Placebo | Group Treatment
Number analyzed (Participants) | 39 | 38
Participants | 12 | 5

5. Secondary Outcome: Inflammatory Processes in the Scalp and Blood Vessels
Description: Signs of inflammation were assessed by trichoscopic evaluation of the scalp and superficial vessels in the target area. The endpoint reflects the proportion of participants with trichoscopic signs consistent with inflammatory processes (scalp inflammation and/or vascular changes) at the specified time point.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Group Placebo | Group Treatment
Number analyzed (Participants) | 39 | 38
Participants | 20 | 6

ADVERSE EVENTS:
Time Frame: "From first dose (Day 1) through end of follow-up (Day 90)."
Description: Adverse events were collected throughout the study period (Day 1-Day 90) via participant reporting and assessment at study visits. Events were recorded by study staff; allergic reactions were monitored due to product ingredients (fish and nuts).
Arm/Group | Group Placebo | Group Treatment
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Placebo (N=40) | Group Treatment (N=40)
Food allergy / allergic reaction (Immune system disorders) | 1 (1) | 1 (1) — Suspected food allergy/allergic reaction - led to discontinuation.

LIMITATIONS AND CAVEATS:
Results are based on participants with available Day 90 assessments (Placebo n=39, Treatment n=38). Three participants did not complete the study (adverse events n=2; lost to follow-up n=1) and were not included in the Day 90 analysis, which may introduce attrition bias and limits generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT06605768/Prot_SAP_000.pdf